CLINICAL TRIAL: NCT01510457
Title: Milnacipran for the Pain, Sensory Sensitization and Mood Changes in Knee Osteoarthritis
Brief Title: Milnacipran for Chronic Pain in Knee Osteoarthritis
Acronym: KOA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Norman Harden (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Dr. Norman Harden, Principal Investigator, Shirley Ryan AbilityLab
Organization: Shirley Ryan AbilityLab (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAV-MD-23
Record Dates: First submitted 2011-11-29; First posted 2012-01-16 (Estimated); Results first posted 2015-01-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-05

CONDITIONS: Knee Osteoarthritis; Degenerative Joint Disease; Chronic Pain
Keywords: Knee Osteoarthritis; Degenerative Joint Disease; Chronic Pain; Knee Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Chronic Pain | interventions — Milnacipran; Tablets; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): BID placebo
  Interventions: Drug: Placebo
- Milnacipran (Experimental): Uptitration from 10mg to 50mg BID Milnacipran
  Interventions: Drug: Milnacipran

INTERVENTIONS:
Drug: Milnacipran — Total target dose of 200 mg/day. Subjects will titrate-up according to the following schedule: 25 mg/d (2 pills, 2 days), 50mg mg/d (4 pills, 2 days), 100mg/d (2 pills, 3 days), 150 mg/d (3 pills, 4 days), and steady state is reached once the study participant ingests 200 mg/d(4 pills). The steady state is maintained for 44 days (approx. 6 weeks). If intolerable side effects occur, the dose may be reduced to last tolerable does, a minimum of 100 mg/day at the discretion of the PI. Subjects unable to tolerate 100 mg/day will be discontinued from the study. A 2-week down-titration will be used.
  Other Names: Savella (milnacipran HCL) Tablets
  Arms: Milnacipran
Drug: Placebo — Subjects will receive identical placebo pills and dosing schedule as that of participants receiving active study medication.
  Other Names: "Sugar Pill"
  Arms: Sugar Pill

SUMMARY:
The patients are asked to take part in this study because you have chronic pain as a result of knee osteoarthritis. This study is done to investigate the pain relieving effects of the study drug Savella (milnacipran HCl) for people who experience chronic osteoarthritis pain. The purpose of this research is to look at how the study drug can be used to benefit people who experience osteoarthritis knee pain. This is a phase IV study done to study the safety and effectiveness of the drug. At this point the drug is already approved by the Food and Drug Administration for people with fibromyalgia but it has not yet been approved for people with knee osteoarthritis.

DETAILED DESCRIPTION:
If you are in this study, you will be placed in one of two study groups: one group will receive the study drug and one will receive a placebo. You will be assigned a study group by chance using a process similar to the flip of a coin.

At the first visit (week one) we will review and sign the informed consent, obtain your medical health history, and conduct a brief physical exam. You will also complete several questionnaires about your pain. You will be assessed for your eligibility to participate in this study. If you are eligible, we will conduct some physical and sensory tests and collect a blood sample. The physical tests include a stair climb, 6-minute treadmill test and a 1-minute sit to stand test. The sensory tests allow us to understand your perception of various stimuli such as vibration, light touch, pinprick, heat, cold, hot pain, and cold pain. At the end of the first visit you will be given an electronic diary to record your pain throughout the study. We will also ask you to wear a device in a T-shirt, similar to an accelerometer, that will be used to record your sleep quality and physical activity for 2 days.

At the second (week two) and third visits (week nine) you will be asked to complete the same questionnaires, physical and sensory tests as during the first visit. You will also have to wear the t-shirt with the device for 2 days after each visit.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain and osteophytes on radiographs OR
* Knee pain plus patient age of 40 years or older, morning stiffness lasting 30 minutes or less, and crepitus (cracking sound) during motion
* Experiences chronic pain for 6 months or longer
* Average pain rating of worse knee is equal to 4 or greater on a 0-10 scale
* If female, is not pregnant or breast feeding, and not currently attempting to conceive; if of childbearing potential, use of a highly effective method of birth control (as determined by Pl)
* Able to walk at least ½ a city block a day, and agrees to try and slowly increase that over the course of study
* Able to read and speak English and provide informed consent
* Able to understand and comply with all data collection methodology including electronic diary
* Subject agrees to 1) continue their stable drug regimen with no changes during the course of study, 2) only use Tylenol 325 mg of tablets (a maximum of 8 tablets a day) for breakthrough pain, and 3) not use Tylenol or any other pain medicines 12 hours before testing.

Exclusion Criteria:

* Subject takes SNRIs (Savella, Cymbalta, Venlafaxine) or other neuroamine re-uptake blockers for mood disorders
* Subject is allergic to SSRIs, SNRIs, or milnacipran
* Subject has severe or untreated psychiatric disturbance (e.g. mania, depression, anxiety, substance dependence)
* Subject is medicated with 'triptans, MAOIs, SSRIs, other SNRIs, tricyclic or heterocyclic antidepressants, lithium, epinephrine, norepinephrine, clonidine or digoxin during the trial
* Subject has a clinical diagnosis of fibromyalgia
* Subject has severe ongoing or unaddressed medical conditions (e.g. Renal or Hepatic disease [creatinine>1.5 ml/dl; AST or ALT> 3x normal limit], uncontrolled hypertension, severe cardiac rate or rhythm disorders, rheumatologic disease (e.g. polymyalgia rheumatica), narrow angle glaucoma, hyponatremia, clotting disorders, uncontrolled seizure disorder or urinary retention)
* Subject has cardiac implants
* Subject has a knee replacement
* Subject plans to start new pain treatments or therapies during the study (e.g. new pain medication, injections, PT, surgery)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Harden, MD, Principal Investigator — Center for Pain Studies, Rehabilitation Institute of Chicago

REFERENCES:
- [Derived] Leaney AA, Lyttle JR, Segan J, Urquhart DM, Cicuttini FM, Chou L, Wluka AE. Antidepressants for hip and knee osteoarthritis. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012157. doi: 10.1002/14651858.CD012157.pub2. PMID 36269595

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Milnacipran
Started | 17 | 29
Completed | 12 | 26
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Milnacipran | Total
Number analyzed (Participants) | 12 | 26 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (7) | 57 (9) | 56 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 23
  Male | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 26 | 38

OUTCOME MEASURES:

1. Primary Outcome: McGill Pain Questionnaire - Short Form
Description: The MPQ-SF is a well-validated pain measure that permits separation of the sensory and affective components of pain, which are added together to compute a total score. The scale ranges from 0-45 (0=no pain, 45=the most pain).
Time Frame: Collected at 2 visits over 11 weeks: Visit 1 and Visit 3.
Measure: Mean (Standard Deviation); unit: units on a pain scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on a pain scale
  MPQ-SF (total) Visit 1 | 10.5 (7.3) | 15.7 (12.2)
  MPQ-SF (total) Visit 3 | 6.0 (5.9) | 12.3 (9.6)

2. Secondary Outcome: Daily Diary Entries With Pain, Fatigue and Functioning Scores Three Times a Day
Description: Averages of daily diary outcomes were taken over the first and last week of the trial (week 1 and week 11) to compare pre and post treatment. diary was filled out 3 times a day and asked subjects to rate pain at rest, pain when walking, and fatigue on a scale 0-10 (0=none, and 10=the worst)
Time Frame: electronic diary entries with pain, fatigue and functioning scores were completed three times a day during week 1 and week 11
Measure: Mean (Standard Deviation); unit: units on a 0-10 NRS scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on a 0-10 NRS scale
  Ave Pain at rest reported on Diary over Week 1 | 4.1 (2.1) | 5.6 (2.1)
  Ave Pain at rest reported on Diary over Week 11 | 2.0 (1.5) | 3.7 (1.9)
  Ave Pain walking reported on Diary over Week 1 | 5.2 (2.0) | 6.4 (2.1)
  Ave Pain walking reported on Diary over Week 11 | 3.1 (1.7) | 4.6 (2.0)
  Ave Fatigue reported on Diary over Week 1 | 4.3 (2.0) | 4.4 (2.8)
  Ave Fatigue reported on Diary over Week 11 | 3.4 (2.4) | 2.8 (1.5)

3. Primary Outcome: PamSys Actigraph Data
Description: We used a body worn sensor (PAMSys™, Biosensics, LLC, MA)(25-27) embedded in a comfortable t-shirt at the sternal level. Participants wore the PAMSys after the visit for 48 hours. The device provides values related to subjects spontaneous physical activity including percentage of time standing and walking. These variables provide different indexes of participants' level of activity and activity organization, and were reported by subjects with KOA pain as relevant.
Time Frame: 48 hours after visit 3
Measure: Mean (Standard Error); unit: percentage of activity (over 48 hours)
Arm/Group | Sugar Pill | Milnacipran
Number analyzed (Participants) | 12 | 26
percentage of activity (over 48 hours)
  percentage of time standing | 18.154 (1.816) | 17.675 (1.218)
  percentage of time walking | 10.218 (1.440) | 11.198 (.966)

4. Primary Outcome: Pain Anxiety Symptoms Scale (PASS)
Description: Anxiety scores were collected at least two data points. The Pain Anxiety Symptoms Scale (PASS) is a scale from 0 - 100, where 0 = no anxiety and 100 = the most anxiety.
Time Frame: Collected at 2 visits over 11 weeks: Visit 1 and Visit 3.
Measure: Mean (Standard Deviation); unit: units on an anxiety scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on an anxiety scale
  PASS-20 (total) Visit 1 | 34.5 (18.6) | 39.1 (23.8)
  PASS-20 (total) Visit 3 | 22.0 (13.7) | 31.2 (22.6)

5. Primary Outcome: Pain Disability Index (PDI)
Description: The PDI is a seven-item, validated instrument that assesses perceived disability in seven key life areas. It provides a total disability score, and is an indirect measure of self efficacy. The Pain Disability Scale is a scale from 0 - 70, where 0 = no Disability and 70 = the most Disability.
Time Frame: Collected at 2 visits over 11 weeks: Visit 1 and Visit 3.
Measure: Mean (Standard Deviation); unit: units on a disability scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on a disability scale
  Pain Disability Index (total)_Visit 1 | 28 (14) | 31 (11)
  Pain Disability Index (total)_Visit 3 | 15 (10) | 26 (18)

6. Primary Outcome: Center for Epidemiological Studies Depression Scale CESD-10 (CES-D 10)
Description: The CES-D 10 is a 10-item questionnaire that has been validated for the assessment of depressive symptomatology. The Depression Scale is a scale with a sum score from 0 - 30, where 0 = no Depression and 30 = the most Depression.
Time Frame: Collected at 2 visits over 11 weeks: Visit 1 and Visit 3.
Measure: Mean (Standard Deviation); unit: units on the depression scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on the depression scale
  CES-D-10 (total) Visit 1 | 7 (5) | 6 (4)
  CES-D-10 (total) Visit 3 | 6 (4) | 9 (7)

7. Primary Outcome: Pain Visual Analogue Scale
Description: Pain Visual Analogue Scale from 0-100 (0= no pain, and 100= most pain).
Time Frame: Collected at 2 visits over 11 weeks: Visit 1 and Visit 3.
Measure: Mean (Standard Deviation); unit: units on a 100mm pain scale
Arm/Group | Milnacipran | Sugar Pill
Number analyzed (Participants) | 26 | 12
units on a 100mm pain scale
  VAS now Visit 1 | 44 (24) | 55 (28)
  VAS now Visit 3 | 20 (22) | 51 (24)

ADVERSE EVENTS:
Arm/Group | Milnacipran | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/12
Other Adverse Events (participants affected / at risk) | 9/26 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=26) | Sugar Pill (N=12)
Nausea (General disorders) | 3 | 0
Fatigue (General disorders) | 3 | 0
Trouble Sleeping (General disorders) | 2 | 0
Constipation (General disorders) | 2 | 0
Headache (General disorders) | 2 | 0
Transient tachycardia (Cardiac disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No